CLINICAL TRIAL: NCT06999460
Title: A Novel Approach to Shoulder Analgesia: Infraspinatus-teres Minor Block for Pre-emptive Analgesia in Patients Undergoing Shoulder Surgeries: A Randomized Controlled Study
Brief Title: Analgesic Effect of Infraspinatus-teres Minor Block for Pre-emptive Analgesia in Patients Undergoing Shoulder Surgeries.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1299
Record Dates: First submitted 2025-05-19; First posted 2025-05-31 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Preemptive Analgesia
Keywords: infraspinatus teres minor block; preemptive analgesia; shoulder surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: To study the efficacy of the infraspinatus-teres minor (ITM) block as pre-emptive analgesia in pain management in patients undergoing shoulder surgeries.
Who Masked: Outcomes Assessor
Masking Description: Anesthetist not sharing in the study will assess outcomes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- *Group Infraspinatus teres minor block (ITM group) (Active Comparator): Patients in this group will receive a unilateral ultrasound-guided Infraspinatus-teres minor (ITM) block with injection of local anesthetics (20 mL of bupivacaine 0.25% (50 mg), 50 mcg dexmedetomidine (0.5 ml) and 8 mg dexamethasone (2 ml)) before induction of general anesthesia
  Interventions: Procedure: Infraspinatus teres minor block group
- Control group (group C) (Active Comparator): Patients in this group will receive general anesthesia.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Infraspinatus teres minor block group — Patients in this group will receive a unilateral ultrasound-guided Infraspinatus-teres minor (ITM) block with injection of local anesthetics (20 mL of bupivacaine 0.25% (50 mg), 50 mcg dexmedetomidine (0.5 ml) and 8 mg dexamethasone (2 ml)) before induction of general anesthesia
  Arms: *Group Infraspinatus teres minor block (ITM group)
Procedure: Control group — Patients in this group will receive general anesthesia
  Arms: Control group (group C)

SUMMARY:
The aim of the study to evaluate the efficacy of the infraspinatus-teres minor (ITM) block in improving pre-emptive analgesia, reducing opioid consumption, and enhancing the overall analgesic effect in patients undergoing shoulder surgeries.

DETAILED DESCRIPTION:
To compare between infraspinatus-teres minor versus control group (GA):

1. To measure analgesic parameters including: the total amount of rescue analgesic consumption (morphine) in the first 24 hours post-operatively in each group, duration of analgesia, and total amount of intraoperative fentanyl consumption and
2. To assess pain score by using numerical rate scale (NRS) at rest (static) and during passive or active movement of shoulder joint (dynamic).
3. To assess discharge time from post anesthesia care unit (PACU).
4. To assess side effects of systemic opioids (constipation, itching, dizziness, nausea and vomiting) and complications of infraspinatus-tere minor block.
5. Patients' satisfaction: The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia).

ELIGIBILITY:
Inclusion Criteria:

* • Patients' acceptance.

  * Age: Adults aged 21-65 years old.
  * BMI: 25-30 kg/m2
  * Sex: both sexes (males or females).
  * Patients undergoing unilateral shoulder surgey under general anesthesia.
  * ASA (American Society of Anesthesiologists) physical status classification I to II.
  * Duration of the surgery < 3hours.

Exclusion Criteria:

* • Patients with contraindications to regional anesthesia (e.g. local or systemic infections, or severe neurological or muscular or bleeding disorders or patient on anticoagulant).

  * Allergy to study medications: bupivacaine or dexamethasone, or dexmedetomidine
  * Patients with severe cardiovascular, respiratory, renal, or hepatic diseases, uncontrolled diabetes , or those undergoing chronic opioid therapy.
  * Psychiatric disorders that hinder informed consent or study participation.
  * history of neurological diseases or conditions that would affect the efficacy of nerve blocks (e.g., neuropathy, spinal cord injury, or history of severe muscle weakness).
  * Patients with nerve injury or disease around the shoulder joint, including thoracic outlet syndrome, Multiple sclerosis, cervical disc disease with ipsilateral radiculopathy, or patients with abnormal sensory or motor function of the upper limb.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
total amount of rescue analgesic consumption | for 24 hours
  To assess the total amount of rescue analgesic consumption in the first 24 hours post-operatively in each group.
total amount of intraoperative supplementary fentanyl consumption. | up to 3 hours
  To measure total amount of intraoperative supplementary fentanyl consumption.

SECONDARY OUTCOMES:
Numerical Rate Scale (NRS) at rest (static) and during passive or active movement of shoulder (dynamic). | 30 minutes after arrival in the post-anesthesia care unit (PACU), 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours postoperatively.
  To assess pain score by using numerical rate scale (NRS) at rest (static) and during passive or active movement of shoulder (dynamic). NRS scale will be explained to all patients as follows: 0= no pain and 10= worst pain.
Time to the first request of rescue analgesia postoperatively | 24 hours postoperative
  To assess the time to the first request of rescue analgesia (morphine) postoperatively
Discharge time from post anesthesia care unit (PACU) | 24 hours
  the time from admission to the post-anesthesia care unit (PACU) till discharge from the PACU when the Aldrete score is ≥9).
To assess side effects of systemic opioids | for 24 hours
  To assess side effects of systemic opioids (constipation, itching, dizziness, nausea & vomiting
the incidence of block -related side effects or complications | for 24 hours
  To assess the incidence of block -related side effects or complications (hematoma, infection or LA toxicity).
patient's satisfaction | for 24 hours
  The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points Likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculity of medicine, Zagazig university, Zagazig, Zagazig, Egypt
  - Faculty of human medicine, Zagazig university, Zagazig, Zagazig

IPD SHARING:
Plan to Share IPD: No